CLINICAL TRIAL: NCT04935437
Title: Implementing a Rehabilitation Program in Patients Recovering From Covid-19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Andreas Asimakos, Principal Investigator, Evangelismos Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-1-2021 22
Record Dates: First submitted 2021-06-01; First posted 2021-06-23 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Rehabilitation
Keywords: Rehabilitation; post COVID-19 sequalae

STUDY DESIGN:
Intervention Model Description: Before and after trial matched cohort trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The patients in this arm will be enrolled in a 2 months supervised rehabilitation program. Evaluation will take place at recruitment time and at the end of the program (2 months).
  Interventions: Other: Supervised rehabilitation program.
- Control (No Intervention): The patients in this arm will not be enrolled in a supervised rehabilitation program. Evaluation will take place at recruitment and at 2 months.

INTERVENTIONS:
Other: Supervised rehabilitation program. — The program includes aerobic exercise, strengthening exercises, physiotherapy, psychological support and dietary advice.
  Arms: Intervention

SUMMARY:
Implementation of a supervised rehabilitation program in patients recovering from COVID-19-infection who suffer from limitations and symptoms due to the disease 6 to 8 weeks from hospital discharge. Patients who have been seriously ill and have been admitted to the ward with high oxygen mixtures or have been admitted to the ICU will be selected primarily. The program includes supervised rehabilitation sessions 2 times a week for 2 months. Patients will be evaluated during recruitment and at the end of the program. Patients who can not attend the program due to logistical/transport issues will be re-evaluated in 2 months and constitute the control population. Investigators hypothesis is that post COVID-19 patients who have persistent symptoms, including fatigue following a supervised rehabilitation program will have fewer symptoms after the end of the program compared to similar patients who do not attend a rehabilitation program.

ELIGIBILITY:
Inclusion Criteria: Candidates for inclusion in the study are:

* Patients recovering from COVID-19 disease AND suffering from persistent limitations (>=1 month) of their physical activity and reduction of their quality of life and associated symptoms including shortness of breath, fatigue, weakness of the upper and lower extremities, post-traumatic stress, pain, etc.
* Priority will be given to patients suffering from more symptoms and disabilities. Patients who might suffer more after COVID-19 disease are:

  1. Patients admitted to the ICU, especially those who were intubated.
  2. Patients who needed high oxygen mixtures (high-flow nasal cannula -HFNC, non-re-breathing mask) as well as those who were older and had prolonged hospitalization.

     -

     Exclusion Criteria:
* Patients who suffer from active disease will not be included until they stop being infectious.
* Patients treated with COVID-19 infection where the main reason for hospitalization was not the virus infection (e.g. due to coronary heart disease, surgery, etc.) will also be excluded.
* Patients suffering from dementia,
* patients with myocarditis
* patients with thromboembolic disease that receive anticoagulants for less than a month
* patients chronically paralyzed,
* patients with paraplegia,
* patients with multiple injuries
* patients with serious orthopedic problems that cause disability
* patients suffering from very serious underlying diseases such as end-stage cancer,
* patients with neurological diseases that cause disability, require rehabilitation clinics and special interventions (speech therapy, kinesiotherapy, patients with tracheostomy etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
Assessment of fatigue with FACIT fatigue Scale | 2 months
  The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued). Score range is from 0-52 and the higher the score the better QOL (quality of life).
Assessment of fatigue using chalder fatigue scale. | 2 months
  The chalder fatigue scale is scored bimodally with a range from 0 to 11 assessing the number of symptoms. It is also scored in Likert style with a range of 0-33 in order to asses the severity of symptoms. The higher the scores indicate more and more severe symptoms.
Assessment of fatigue with Fatigue Severity Scale | 2 months
  Assessment of fatigue using the Fatigue Severity Scale. The minimum score is 9 and maximum score is 63. Higher values mean higher fatigue severity.
Assessment of respiratory symptoms after COVID-19 with CAT. | 2 months
  Assessment of symptoms after COVID-19 using the COPD Assessment Test (CAT). Minimum score is 0 and maximum score is 40. Patients with higher scores are more impaired. Patients with a score of 10 or more are considered significantly impaired after COVID-19 infection.

SECONDARY OUTCOMES:
Assessment of quality of life using SF-36 questionnaire. | 2 months
  The RAND 36-Item Health Survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Assessment of shortness of breath | 2 months
  Assessment of shortness of breath using the modified MRC scale. The minimum score is 0 and maximum score is 4. Higher values mean more dyspnea.
Assessment of functional capacity with 6MWT. | 2 months
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Assessment of symptoms after COVID-19 with PCFS. | 2 months
  Assessment of symptoms after COVID-19 using the Post-COVID-19 Functional Status scale (PCFSS). Minimum score is 0 and maximum score is 4. Patients with higher scores are more impaired. Patients with a score of 2 or more are considered significantly impaired after COVID-19 infection.
Assessment of lower extremity strength | 2 months.
  Assessment of lower extremity strength using a dynamometer.
Assessment of functional capacity with one minute sit to stand test. | 2 months
  The one minute sit to stand test assesses functional lower extremity strength, transitional movements, balance, and fall risk.The 1-minute STS test is performed with a chair of standard height of 46 cm without arm rests. The patient is ensured to be seated upright on the chair positioned against a wall. The patient sits with the knees and hips flexed to 90°, feet placed flat on the floor hip-width apart, and the hands placed on the hips. Every get up from the chair is validated to check if complete sit-to-stand-to-sit sequence is achieved. The number of repetitions is measured.
Assessment of functional capacity with Short Physical Performance Battery. | 2 months
  Short Physical Performance Battery is a simple test to measure lower extremity function using tasks that mimic daily activities. The SPPB examines 3 areas of lower extremity function; static balance, gait speed, and getting in and out of a chair. SPPB scores range from zero to 12 possible points, a score lower than 10 indicates one or more mobility limitations
Assessment of Post Traumatic Stress Disorder with the Impact of Event Scale revised. | 2 months
  The Impact of Event Scale - Revised (IES-R) is designed as a measure of post-traumatic stress disorder (PTSD) symptoms. It's a 22-item self report measure that assesses subjective distress caused by traumatic events. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score (ranging from 0 to 88) and subscale scores can also be calculated for the Intrusion, Avoidance, and Hyperarousal subscales.
Assessment of anxiety and depression with HADS | 2 months
  The Hospital Anxiety and Depression Scale (HADS) measures anxiety and depression in a general medical population of patients. HADS focuses on non-physical symptoms so that it can be used to diagnose depression and/or anxiety in people with significant physical ill-health.The questionnaire comprises seven questions for anxiety and seven questions for depression.
  For both scales, scores of less than 7 indicate non-cases 8-10 Mild 11-14 Moderate 15-21 Severe
Assessment of lung diffusion capacity. | 2 months
  Assessment of lung diffusion capacity through measurement of diffusing capacity of the lung for carbon monoxide (CO) (DLCO)
Assessment of respiratory function with FVC | 2 months
  Assessment of respiratory function measuring Forced Vital Capacity with spirometry.
Assessment of quality of life using EQ-5D-5L questionnaire. | 2 months
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Assessment of physical activity with IPAQ. | 2 months
  International Physical Activity Questionnaire (IPAQ) is 27 item self report measure of physical activity for adults 15 to 69 years old. There two forms of output from scoring the IPAQ, in categories (low, moderate and high activity), or as continuous variables as MET minutes per week. MET minutes represent the amount of energy expended carrying out physical activity. The higher the score the more active the participant.
Assessment of balance. | 2 months
  The Activities-Specific Balance Confidence (ABC) scale is used. Patients give their answers in % of confidence and score ranges from 0% (worst possible balance confidence) to 100% .
Assessment of respiratory function with FEV1 | 2 months
  Assessment of respiratory function measuring Forced Expiratory Volume in 1 minute with spirometry.
Assessment of cognitive dysfunction | 2 months
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment. The MoCA test is a one-page 30-point test, scores range between 0 and 30. A score of 26 or over is considered to be normal.
Assessment of depression with Beck Depression Inventory | 2 months
  The Beck Depression Inventory (BDI, BDI-1A, BDI-II), is a 21-question multiple-choice self-report inventory for measuring the severity of depression.
  When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores were as follows:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression. Higher total scores indicate more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelismos Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spruit MA, Holland AE, Singh SJ, Tonia T, Wilson KC, Troosters T. COVID-19: interim guidance on rehabilitation in the hospital and post-hospital phase from a European Respiratory Society- and American Thoracic Society-coordinated international task force. Eur Respir J. 2020 Dec 3;56(6):2002197. doi: 10.1183/13993003.02197-2020. Print 2020 Dec. PMID 32817258
- [Background] Sally Singh, Charlotte Bolton, Claire Nolan, Theresa Harvey-Dunstan, Bronwen Connolly, William Man and Paul Walker. Delivering rehabilitation to patients surviving COVID-19 using an adapted pulmonary rehabilitation approach - BTS guidance [Internet]. British Thoracic Society; 2020. Available from: https://www.brit-thoracic.org.uk/document-library/quality-improvement/covid-19/pulmonary-rehabilitation-for-covid-19-patients/
- [Background] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Background] Daynes E, Gerlis C, Briggs-Price S, Jones P, Singh SJ. COPD assessment test for the evaluation of COVID-19 symptoms. Thorax. 2021 Feb;76(2):185-187. doi: 10.1136/thoraxjnl-2020-215916. Epub 2020 Nov 4. PMID 33148809
- [Background] Klok FA, Boon GJAM, Barco S, Endres M, Geelhoed JJM, Knauss S, Rezek SA, Spruit MA, Vehreschild J, Siegerink B. The Post-COVID-19 Functional Status scale: a tool to measure functional status over time after COVID-19. Eur Respir J. 2020 Jul 2;56(1):2001494. doi: 10.1183/13993003.01494-2020. Print 2020 Jul. PMID 32398306